CLINICAL TRIAL: NCT00839293
Title: Comparison of Fenofibric Acid Bioavailability From 45 mg and 135 mg Strength ABT-335 Capsules
Brief Title: Comparison of Fenofibric Acid Bioavailability From ABT-335 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Maureen Kelly, MD/Senior Medical Director, Abbott
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M10-788
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Bioavailability
MeSH Terms: interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; fenofibric acid; Fenofibrate

ARMS (2):
- A (Experimental): ABT -335 capsules 135mg
  Interventions: Drug: ABT-335
- B (Experimental): ABT-335 capsules 45mg
  Interventions: Drug: ABT-335

INTERVENTIONS:
Drug: ABT-335 — Once, see arm description for more information
  Other Names: fenofibric acid; Trilipix

SUMMARY:
The purpose of this study is to evaluate the safety and compare the bioavailability of fenofibric acid from 2 different dosage strengths of ABT-335.

ELIGIBILITY:
Inclusion Criteria:

* A condition of general good health
* BMI 18 to 29

Exclusion Criteria:

* Currently enrolled in another clinical study
* Females who are pregnant or breast-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the bioavailability of ABT-335 in healthy subjects as measured by timed pharmacokinetic blood draws from pre-dose (0 hour) to 120 hours post dose | 14 Days
To evaluate the safety and tolerability of ABT-335 in healthy adults after single dosage | 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Kelly, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 16862, Waukegan, Illinois, United States